CLINICAL TRIAL: NCT03787732
Title: Preventing Cardiovascular Collapse With Administration of Fluid Resuscitation During Induction and Intubation (PREPARE II Trial)
Brief Title: Preventing Cardiovascular Collapse With Administration of Fluid Resuscitation During Induction and Intubation
Acronym: PREPARE II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Matthew Semler, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB# 181690
Record Dates: First submitted 2018-12-22; First posted 2018-12-26 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Acute Respiratory Failure; Intubation Complication; Hypotension on Induction
Keywords: Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid Bolus (Active Comparator): For patients randomized to fluid bolus administration, the bedside nurse will obtain 500 mL of a crystalloid solution of the operator's choosing, connect this volume to intravenous infusion tubing, and attach the tubing to any intravenous catheter or intraosseous device. The crystalloid solution will then be placed above the level of the intravenous or intraosseous device and allowed to infuse by gravity or pressure bag. At any time after the initiation of fluid bolus administration, the operator can choose to begin the procedure by administering sedation. Fluid loading will continue until all 500 mL are infused. Fluid infusing prior to the decision to perform endotracheal intubation will not be altered by the current study.
  Interventions: Drug: Fluid Bolus
- No Fluid Bolus (Active Comparator): For patients randomized to no fluid bolus administration, no additional intravenous crystalloid administration will be initiated between randomization and two minutes after completion of endotracheal intubation. Fluid infusing prior to the decision to perform endotracheal intubation will not be affected by the study. Treating clinicians may initiate a fluid bolus at any time for the treatment of cardiovascular collapse (not considered a protocol violation). Treating clinicians may also initiate a fluid bolus at any time if felt to be mandatory for the safe treatment of the patient (if between randomization and two minutes after intubation and in the absence of cardiovascular collapse this will be recorded as a protocol violation).
  Interventions: Other: No Fluid Bolus

INTERVENTIONS:
Drug: Fluid Bolus — 500 milliliters of an intravenous crystalloid solution of the operator's choosing
  Other Names: intravenous crystalloid fluid, 500 mL
  Arms: Fluid Bolus
Other: No Fluid Bolus — No additional intravenous crystalloid administration initiated between randomization and two minutes after completion of endotracheal intubation
  Arms: No Fluid Bolus

SUMMARY:
Complications are common during tracheal intubation of critically ill patients. Nearly one in five patients undergoing intubation in the intensive care unit experiences cardiovascular collapse, defined as severe hypotension, vasopressor administration, cardiac arrest or death. Cardiovascular collapse during intubation is associated with increased resource utilization and decreased survival. Administration of 500 mL of intravenous crystalloid solution beginning prior to induction may prevent cardiovascular collapse. The only prior trial examining fluid bolus administration during intubation found no effect on cardiovascular collapse or clinical outcomes overall, but a hypothesis-generating subgroup analysis suggested potential benefit to fluid bolus administration among patients receiving positive pressure ventilation between induction and laryngoscopy. Therefore, we propose a randomized trial comparing fluid bolus administration versus none with regard to cardiovascular collapse among critically adults undergoing intubation with positive pressure ventilation between induction and laryngoscopy.

DETAILED DESCRIPTION:
The PREPARE II trial is a prospective, parallel group, pragmatic, randomized trial comparing the effect of a preintubation fluid bolus to no preintubation fluid bolus on the incidence of cardiovascular collapse during and after endotracheal intubation in critically ill adults.

Patients admitted to the study units who are deemed by their clinical team to require intubation and fulfill inclusion criteria without meeting exclusion criteria will be randomized 1:1 to receive either an intravenous fluid bolus or no intravenous fluid bolus. All other decisions regarding airway management will remain at the discretion of the treating provider.

Conduct of the trial will be overseen by a Data Safety Monitoring Board. An interim analysis will be performed after the enrollment of 375 patients. The analysis of the trial will be conducted in accordance with a pre-specified statistical analysis plan, which will be submitted for publication or made publicly available prior to the conclusion of enrollment.

The primary outcome is cardiovascular collapse - a composite endpoint defined as one or more of the following:

1. Death within 1 hour of intubation
2. Cardiac arrest within 1 hour of intubation
3. New systolic blood pressure < 65 mmHg between induction and 2 minutes after completion of intubation
4. New or increased vasopressor receipt between induction and 2 minutes after completion of intubation

The secondary outcome is 28-day in-hospital mortality

ELIGIBILITY:
Inclusion Criteria:

1. Patient is undergoing endotracheal intubation in a participating unit
2. Planned operator is a provider expected to routinely perform endotracheal intubation in the participating unit
3. Patient is at least 18 years of age
4. Administration of sedation is planned (with or without neuromuscular blockade)
5. Positive pressure ventilation between induction and laryngoscopy is planned (e.g., non-invasive ventilation or bag-mask ventilation)

Exclusion Criteria:

1. Prisoners
2. Pregnant patients
3. Urgency of intubation precludes safe performance of study procedures
4. Operator feels administration of a fluid bolus is indicated or contraindicated for the safe performance of the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1067 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Cardiovascular collapse | 1 hour
  A composite endpoint defined as one or more of the following
  * New systolic blood pressure < 65 mmHg between induction and 2 minutes after intubation
  * New or increased vasopressor between induction and 2 minutes after intubation
  * Cardiac arrest within 1 hour of intubation
  * Death within 1 hour of intubation

SECONDARY OUTCOMES:
28-day in-hospital mortality | 28 days

OTHER OUTCOMES:
New systolic blood pressure < 65 mmHg between induction and 2 minutes after intubation | from induction to 2 minutes following tracheal intubation
New or increased vasopressor between induction and 2 minutes after intubation | from induction to 2 minutes following tracheal intubation
Cardiac arrest within 1 hour of intubation | 1 hour
Death within 1 hour of intubation | 1 hour
Lowest systolic blood pressure between induction and 2 minutes after intubation | from induction to 2 minutes following tracheal intubation
Change in systolic blood pressure from induction to lowest systolic blood pressure | between induction and 2 minutes following procedure
Ventilator-free days | 28 days
ICU-free days | 28 days
Lowest oxygen saturation | from induction to 2 minutes following tracheal intubation
  Lowest arterial oxygen saturation between induction and 2 minutes after intubation
Incidence of hypoxemia | from induction to 2 minutes following tracheal intubation
  Incidence of oxygen saturation < 90% between induction and 2 minutes after intubation
Incidence of severe hypoxemia | from induction to 2 minutes following tracheal intubation
  Incidence of oxygen saturation < 80% between induction and 2 minutes after intubation
Oxygen saturation at 24 hours after intubation | 24 hours
Fraction of inspired oxygen at 24 hours after intubation | 24 hours
Positive end expiratory pressure at 24 hours after intubation | 24 hours
Systolic blood pressure at 24 hours after intubation | 24 hours
Additional intravenous fluids initiated between induction and 2 minutes after intubation | from induction to 2 minutes following tracheal intubation
Time from induction to successful intubation | Duration of procedure (minutes)
Cormack-Lehane grade of glottic view on first attempt | Duration of procedure (minutes)
Difficulty of intubation | Duration of procedure (minutes)
  Operator-reported difficulty of intubation on a three-point ordinal scale of: easy, moderate, or difficult.
Incidence of successful intubation on the first laryngoscopy attempt | Duration of procedure (minutes)
Number of laryngoscopy attempts | Duration of procedure (minutes)
Need for additional airway equipment or a second operator | Duration of procedure (minutes)

CONTACTS AND LOCATIONS:
Overall Officials: David R Janz, MD, MSCI, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans; Derek W Russell, MD, Principal Investigator — University of Alabama at Birmingham
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - Ochsner Medical Center | Ochsner Health System, New Orleans, Louisiana
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Russell DW, Casey JD, Gibbs KW, Ghamande S, Dargin JM, Vonderhaar DJ, Joffe AM, Khan A, Prekker ME, Brewer JM, Dutta S, Landsperger JS, White HD, Robison SW, Wozniak JM, Stempek S, Barnes CR, Krol OF, Arroliga AC, Lat T, Gandotra S, Gulati S, Bentov I, Walters AM, Dischert KM, Nonas S, Driver BE, Wang L, Lindsell CJ, Self WH, Rice TW, Janz DR, Semler MW; PREPARE II Investigators and the Pragmatic Critical Care Research Group. Effect of Fluid Bolus Administration on Cardiovascular Collapse Among Critically Ill Patients Undergoing Tracheal Intubation: A Randomized Clinical Trial. JAMA. 2022 Jul 19;328(3):270-279. doi: 10.1001/jama.2022.9792. PMID 35707974
- [Derived] Russell DW, Casey JD, Gibbs KW, Dargin JM, Vonderhaar DJ, Joffe AM, Ghamande S, Khan A, Dutta S, Landsperger JS, Robison SW, Bentov I, Wozniak JM, Stempek S, White HD, Krol OF, Prekker ME, Driver BE, Brewer JM, Wang L, Lindsell CJ, Self WH, Rice TW, Semler MW, Janz D; PREPARE II Investigators. Protocol and statistical analysis plan for the PREventing cardiovascular collaPse with Administration of fluid REsuscitation during Induction and Intubation (PREPARE II) randomised clinical trial. BMJ Open. 2020 Sep 18;10(9):e036671. doi: 10.1136/bmjopen-2019-036671. PMID 32948554